CLINICAL TRIAL: NCT01225289
Title: The Study of the Effects of Vitamin A Supplementation on Immune System and Th1/Th2 Balance in Patients With Multiple Sclerosis
Brief Title: Impact of Vitamin A Supplementation on Immune System in Multiple Sclerosis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ali Akbar Saboor Yaraghi, Assistant Professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 88-03-27-9576
Record Dates: First submitted 2010-09-06; First posted 2010-10-21 (Estimated); Results first posted 2014-03-14 (Estimated); Last update posted 2014-03-14 (Estimated); Status verified 2014-02

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Vitamin A; CD4-Positive T-Lymphocytes; Th1 Cells; Th2 Cells
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Vitamin A; retinol palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- with Multiple Sclerosis/ vitamin A (Active Comparator): Patients with MS confirmed Relapsing Remitting Type who receive 25000 IU/day vitamin A
  Interventions: Dietary Supplement: Vitamin A
- with Multiple Sclerosis/ placebo (Placebo Comparator): Patients with Multiple Sclerosis confirmed Relapsing Remitting Type who receive 1 cap of placebo per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin A — 25000 IU/day (one capsule per day) Vitamin A for 6 months
  Other Names: Retinyl palmitate
  Arms: with Multiple Sclerosis/ vitamin A
Drug: Placebo — 1 capsule per day for six months
  Arms: with Multiple Sclerosis/ placebo

SUMMARY:
The aim of this study is to study the comparison between the effects of supplementation with 25000 IU preformed vitamin A (retinyl palmitate) or placebo for 6 months on immune system and Th1/Th2 balance in patients with Multiple Sclerosis.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic inflammatory disease where Th1 like responses from myelin-specific CD4+ T cells, as secretion of pro-inflammatory IFN-g, are believed to play a major role in the pathogenesis. The myelin-specific T cells that mediate tissue destruction in MS are believed to become activated outside the central nervous system (CNS) in lymphoid tissue and when they cross the blood brain barrier they will re-encounter their antigen. Immune deviation is the redirection of the immune response from most often Th1 like responses to Th2 like responses, even though the opposite can also occur. Vitamin A (VA) or VA-like analogs known as retinoids, are potent hormonal modifiers of type 1 or type 2 responses but a definitive description of their mechanism(s) of action is lacking. High level dietary vitamin A enhances Th2 cytokine production and IgA responses, and is likely to decrease Th1 cytokine production. Retinoic acid inhibits IL 12 production in activated macrophages, and RA pretreatment of macrophages reduces IFNγ production and increases IL4 production in antigen primed CD4 T cells. Supplemental treatment with vitamin A or retinoic acid (RA) decreases IFNγ and increases IL5, IL10, and IL4 production. Thus, vitamin A deficiency biases the immune response in a Th1 direction, whereas high level dietary vitamin A may bias the response in a Th2 direction.

ELIGIBILITY:
Inclusion Criteria:

Patients who have used interferon beta in last 3 months. Patients with 1-5 EDSS

Exclusion Criteria:

* Patients who have diseases which affect on Th1/Th2 balance such as asthma, active viral infections, and autoimmune diseases, OR
* Patients who have allergy to vitamin A compounds, OR
* Patients who have used vitamin supplements in last 3 months.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-10; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali Akbar Saboor Yaraghi, PhD, Principal Investigator — Tehran University of Medical Sciences; Sima Jafarirad, PhD student, Principal Investigator — Tehran University of Medical Sciences
Locations (2):
- Iran (2):
  - Tehran University of Medical Sciences, School of Public Health Tehran, Tehran, Iran, Islamic Republic o, Tehran, Tehran Province
  - Tehran University of Medical Sciences, School of Public Health, Tehran, Tehran Province

REFERENCES:
- [Derived] Mohammadzadeh Honarvar N, Harirchian MH, Koohdani F, Siassi F, Abdolahi M, Bitarafan S, Salehi E, Sahraian MA, Eshraghian MR, Saboor-Yarghi AA. The effect of vitamin A supplementation on retinoic acid-related orphan receptor gammat (RORgammat) and interleukin-17 (IL-17) gene expression in Avonex-treated multiple sclerotic patients. J Mol Neurosci. 2013 Nov;51(3):749-53. doi: 10.1007/s12031-013-0058-9. Epub 2013 Jul 19. PMID 23868508

RESULTS

PARTICIPANT FLOW:
Groups:
- With Multiple Sclerosis/ Placebo: Patients with Multiple Sclerosis confirmed Relapsing Remitting Type who receive 1 cap of placebo/day
Period: Overall Study
Arm/Group | With Multiple Sclerosis/ Vitamin A | With Multiple Sclerosis/ Placebo
Started | 18 | 18
Completed | 18 | 17
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | With Multiple Sclerosis/ Vitamin A | With Multiple Sclerosis/ Placebo | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 35
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.22 (7.26) | 31.05 (5.94) | 32.17 (6.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  Iran, Islamic Republic of | 18 | 17 | 35

OUTCOME MEASURES:

1. Primary Outcome: Difference Serum Levels of High-sensitive C-reactive Protein (Hs-CRP), Before and After of Supplementation
Time Frame: first day and after 6 month
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | With Multiple Sclerosis/ Vitamin A | With Multiple Sclerosis/ Placebo
Number analyzed (Participants) | 18 | 17
mg/L | 1.2 (0.5) | -0.6 (0.4)
Statistical Analysis 1: Comparison: With Multiple Sclerosis/ Vitamin A vs With Multiple Sclerosis/ Placebo; Test type: Superiority or Other; p < 0.01, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Difference of IL-4 Levels in Supernatant of Peripheral Blood Mononucleated Cells (PBMCs) Stimulated With Phytohemagglutinin (PHA), Before and After of Supplementation
Time Frame: first day and after 6 month
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | With Multiple Sclerosis/ Vitamin A | With Multiple Sclerosis/ Placebo
Number analyzed (Participants) | 18 | 17
pg/ml | 2.5 (1.2) | 1.5 (1)

3. Secondary Outcome: Difference of Retinol Binding Protein (RBP) / Transthyretin (TTR) Ratio, (Difference of RBP/ TTR Ratio), Before and After of Supplementation
Time Frame: first day and after 6 month
Measure: Mean (Standard Error); unit: ratio
Arm/Group | With Multiple Sclerosis/ Vitamin A | With Multiple Sclerosis/ Placebo
Number analyzed (Participants) | 18 | 17
ratio | 0.2 (0.2) | -0.4 (0.5)

4. Secondary Outcome: Peripheral Blood Mononucleated Cells (PBMCs) Proliferation Assay (BrdU Colorimetric)
Description: difference of PBMCs proliferation stimulated with myelin oligodendrocyte glycoprotein (MOG), before and after of supplementation
Time Frame: first day and after 6 month
Measure: Mean (Standard Error); unit: absorbance units
Arm/Group | With Multiple Sclerosis/ Vitamin A | With Multiple Sclerosis/ Placebo
Number analyzed (Participants) | 18 | 17
absorbance units | -0.06 (0.08) | -0.13 (0.09)

ADVERSE EVENTS:
Arm/Group | With Multiple Sclerosis/ Vitamin A | With Multiple Sclerosis/ Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 1/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | With Multiple Sclerosis/ Vitamin A (N=18) | With Multiple Sclerosis/ Placebo (N=17)
MS relapsing (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No